CLINICAL TRIAL: NCT05983445
Title: Safety & Efficacy of Genakumab in Patients With Frequent Flares
Brief Title: Safety & Efffficacy of Genakumab in Patients With Frequent Flares
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci048-301
Record Dates: First submitted 2022-12-20; First posted 2023-08-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Acute Gout Arthritis
Keywords: Acute Gout Arthritis
MeSH Terms: interventions — betamethasone dipropionate, betamethasone sodium phosphate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Genakumab (Experimental): Genakumab 200mg s.c
  Interventions: Drug: genakumab; Drug: placebo for Diprospan
- Diprospan (Active Comparator): Diprospan 7mg im
  Interventions: Drug: placebo for genakumab; Drug: Diprospan

INTERVENTIONS:
Drug: genakumab — 200mg s.c.
  Other Names: • Gensci048
  Arms: Genakumab
Drug: placebo for Diprospan — i.m.
  Arms: Genakumab
Drug: placebo for genakumab — s.c.
  Arms: Diprospan
Drug: Diprospan — 7mg i.m.
  Arms: Diprospan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Genakumab Injection in patients with Gouty Arthritis (GA).

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, double-dummy, active-controlled study was to demonstrate the efficacy of Genakumab versus compound betamethasone injection in adult patients with frequent gouty arthritis attacks in whom non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine are contraindicated, are not tolerated, or do not provide an adequate response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years ≤ age ≤75 years
* BMI≤40kg/m2
* Meeting ACR 2015 preliminary criteria for the classification of acute arthritis of primary gout.
* Start of acute gout flare within 4 days prior to enrolled
* History of ≥ 2 gout flares within the 12 months prior to study start
* Evidence of contraindication (absolute or relative), or intolerance, or lack of efficacy for either NSAIDs and/or colchicines
* Baseline pain intensity ≥ 50 mm on the 0-100 mm visual analog scale (VAS)

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
The change in the gout pain intensity in the target joint measured by VAS | 72 hours post-dose
  The Visual Analog Scale (VAS) is an instrument used to measure a person's subjective quantitative evaluation of an item such as pain intensity. In this study patients scored their pain intensity in the joint most affected at Baseline on a 0-100 mm VAS, ranging from no pain (0mm) to unbearable pain (100mm), at 72 hours post-dose. Scores on the 100 mm linear scale were measured to the nearest millimeter from the left.
Time to first new flare | 12 weeks

SECONDARY OUTCOMES:
Patients assessment of gout pain intensity in the target joints measured by VAS(0-100mm) | At 6, 24, 48, and 72 hours and 7 days post-dose
The change in the gout pain intensity in the target joint measured by VAS. | At 6, 24, 48, and 72 hours and 7 days post-dose
The number of patients with at least 1 new gout flare | 12 weeks, 24 weeks, 48 weeks
Time to at Least a 50% Reduction in Baseline Pain Intensity | 7 days
Percent Patients Who Took Rescue Medication | 24 weeks,48 weeks
Time to first flare | 24 weeks, 48 weeks
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | 24weeks, 48weeks
Immunogenicity The incidence of anti-drug antibodies (ADA) and the incidence of neutralizing antibody | 24 weeks, 48 weeks
Genakumab Pharmacokinetics (PK) Serum Concentration During the Treatment Period | 2 hours pre-dose, Days 4，8，29，57，85，169，253 days post-dose
  Blood was collected for Ganakumab levels at2 hours pre-dose, Days 4，8，29，57，85，169，253 days post-dose.

OTHER OUTCOMES:
High Sensitivity C-reactive Protein (hsCRP) | 72 hours, 7 days and 4 weeks post-dose
SF-36 | 8 weeks, 24 weeks and 48 weeks
  The SF-36 measures the impact of disease on overall quality of life (QoL). This 36-item survey has 8 subscales that can be aggregated into physical- and mental-component summary scores. Scores are standardized with the use of norm-based methods based on an assessment of the general U.S. population free of chronic conditions. Scores range from 1-100 with a mean=50 and a standard deviation=10. A higher score indicates less impact on QoL. A negative change score indicates improvement. An ANCOVA model was used with treatment group and baseline SF-36 physical function subscore as covariates.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided